CLINICAL TRIAL: NCT05202600
Title: Justification of Incidental Appendectomy With Respect to Pathohistological Findings
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ognjen Barcot, Ass. Prof., University Hospital of Split
Other Study IDs: KOLO_2022_001
Record Dates: First submitted 2022-01-11; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Appendix Tumor
MeSH Terms: conditions — Appendiceal Neoplasms | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incidental appendectomy (IA): Group IA will include adult patients operated on for colon tumors who have data on age, sex, data on a previously diagnosed colon tumor, data on incidental appendectomy, and a PHD finding for a removed vermiform appendix.
  Interventions: Procedure: Appendectomy
- Acute appendectomy (AA): Group AA will include adult patients who have been operated due to clinical suspicion of acute appendicitis and have data on age, sex, data on the diagnosis of acute appendicitis and accompanying PHD findings of the performed appendectomy.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Surgical removal of the vermiform appendix.
  Other Names: Appendicectomy

SUMMARY:
This study seeks to justify performing an incidental appendectomy according to the following hypotheses:

1. The frequency of neoplasms in pathohistological (PHD) findings of incidental appendectomy (IA) is significantly higher than in PHD findings in appendectomies for acute appendcitis (AA)
2. The number needed to treat (NNT) for appendiceal tumors in the elderly is less than 500.
3. The rate of complicated AA in the elderly population is significantly higher than in the younger age group
4. NNT IA for complicated appendicitis in the elderly is less than 300.
5. NNT IA for potential death due to AA in the elderly is less than 500.

DETAILED DESCRIPTION:
A retrospective cross-sectional study will be done. The archive of all PHD findings will be searched, and then the relevant medical histories at the Clinic of Surgery, University Hospital Center Split in the period from 01.01.2017. to 31.12.2021. The data collection will be done in the period from 01.02.2022. to 31.03.2022. The data collection (extraction) will be done by the main researcher (graduate, Ante Tavra) with at least two other colleagues from the Department of Abdominal-Coloproctological Surgery, University Hospital Center Split (Damir Quien, MD and Dora Bjelanović, MD).

Data will be collected directly from medical history and entered into an overview table. The identity of the respondents will remain secret, and the respondents will be marked exclusively with an identification number. This type of research does not require the informed consent of the patient, and all data collected will be kept in accordance with the provisions of Annex 2 of the Application to Institutional advisory board of UHC Split (approval pending).

ELIGIBILITY:
Inclusion Criteria:

Adult patients operated for colon tumors who have data on age, sex, data on a previously diagnosed colon tumor, data on incidental appendectomy, and a PHD finding for a removed appendix. Adult patients who have been diagnosed with acute appendicitis and have data on age, sex, data on the diagnosis of acute appendicitis and accompanying PHD findings, newly performed appendectomies.

Exclusion Criteria:

We will exclude from the analysis patients who had previous appendectomy, appendectomy has not been performed or we do not have an accompanying PHD finding of the appendix, and patients younger than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients operated in UHC Split Surgery Clinic for colon cancer or acute appendicitis during 5-year period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of appendiceal neoplasms | 01.01.2017. - 31.12.2021.
  Incidence of appendiceal neoplasms in IA which will be compared to the incidence of appendiceal neoplasms AA from respective PH samples.
NNT of IA for the appendiceal neoplasm | 01.01.2017. - 31.12.2021.
  The number of needed incidental appendectomies necessary to avoid one occurence of appendiceal neoplasm

SECONDARY OUTCOMES:
Incidence of complicated appendicits | 01.01.2017. - 31.12.2021.
  Comparison of incidences of complicated appendicits in young vs elderly
NNT of IA for the complicated appendicits in elderly | 01.01.2017. - 31.12.2021.
  The number of needed incidental appendectomies necessary to avoid one occurence of complicated appendicitis in elderly
NNT of IA for the death due to appendicits in elderly | 01.01.2017. - 31.12.2021.
  The number of needed incidental appendectomies necessary to avoid one death from complicated appendicitis in elderly

OTHER OUTCOMES:
Size of the appendix as a predictor of neoplasm | 01.01.2017. - 31.12.2021.
  Receiver operating curve analysis of the size of the vermiform appendix impacting the classification to neoplastic appendix
Definition of the elderly group for appendiceal neoplasm | 01.01.2017. - 31.12.2021.
  Receiver operating curve analysis of the age of the patient impacting the classification to neoplastic appendix
Definition of the elderly group for the complicated appendicitis or death | 01.01.2017. - 31.12.2021.
  Receiver operating curve analysis of the age of the patient impacting the classification to the complicated appendicitis or death

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Barcot, MD, PhD, Principal Investigator — Department of surgery, University Hospital Split
Locations (1):
- University Hospital Split, Split, Split-Dalmatia County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available upon reasonable request by the corresponding author (Ognjen Barcot).

REFERENCES:
- [Result] Akbulut S, Koc C, Sarici B, Ozcan M, Samdanci E, Yilmaz S. Histopathological features of incidental appendectomy specimens obtained from living liver donors. Turk J Gastroenterol. 2020 Mar;31(3):257-263. doi: 10.5152/tjg.2020.19010. PMID 32343238
- [Result] Choksuwattanasakul M. Incidental appendectomy during mini incision post-partum sterilization (Chokchai technique): A prospective cross-sectional study. J Obstet Gynaecol Res. 2017 Dec;43(12):1863-1869. doi: 10.1111/jog.13458. Epub 2017 Sep 11. PMID 28892212
- [Result] Lohsiriwat V, Vongjirad A, Lohsiriwat D. Incidence of synchronous appendiceal neoplasm in patients with colorectal cancer and its clinical significance. World J Surg Oncol. 2009 Jun 2;7:51. doi: 10.1186/1477-7819-7-51. PMID 19490638
- [Result] Huttenbrink C, Hatiboglu G, Simpfendorfer T, Radtke JP, Becker R, Teber D, Hadaschik B, Pahernik S, Hohenfellner M. Incidental appendectomy during robotic laparoscopic prostatectomy-safe and worth to perform? Langenbecks Arch Surg. 2018 Mar;403(2):265-269. doi: 10.1007/s00423-017-1630-5. Epub 2017 Nov 2. PMID 29098385
- [Result] Akbulut S, Koc C, Kocaaslan H, Gonultas F, Samdanci E, Yologlu S, Yilmaz S. Comparison of clinical and histopathological features of patients who underwent incidental or emergency appendectomy. World J Gastrointest Surg. 2019 Jan 27;11(1):19-26. doi: 10.4240/wjgs.v11.i1.19. PMID 30705736
- [Result] McCusker ME, Cote TR, Clegg LX, Sobin LH. Primary malignant neoplasms of the appendix: a population-based study from the surveillance, epidemiology and end-results program, 1973-1998. Cancer. 2002 Jun 15;94(12):3307-12. doi: 10.1002/cncr.10589. PMID 12115365
- [Result] Segev L, Keidar A, Schrier I, Rayman S, Wasserberg N, Sadot E. Acute appendicitis in the elderly in the twenty-first century. J Gastrointest Surg. 2015 Apr;19(4):730-5. doi: 10.1007/s11605-014-2716-9. Epub 2015 Feb 14. PMID 25681217
- [Result] Ahmed HO, Muhedin R, Boujan A, Aziz AHS, Abdulla AM, Hardi RA, Abdulla AA, Sidiq TA. A five-year longitudinal observational study in morbidity and mortality of negative appendectomy in Sulaimani teaching Hospital/Kurdistan Region/Iraq. Sci Rep. 2020 Feb 6;10(1):2028. doi: 10.1038/s41598-020-58847-1. PMID 32029830